CLINICAL TRIAL: NCT03903991
Title: Evaluation of the Reliability of Oesophageal Temperature in THOracic Surgery
Acronym: ThoTem
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18-ThoTem; 2019-A00407-50 (Other: IdRCB)
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypothermia; Thoracic Neoplasm; Anesthesia
Keywords: Thoracic surgery; Body temperature
MeSH Terms: conditions — Hypothermia; Thoracic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracotomy: All patients needing pulmonary surgery under thoracotomy
  Interventions: Other: Temperature recording

INTERVENTIONS:
Other: Temperature recording — Tympanic and oesophageal temperatures will be recorded during the procedure

SUMMARY:
Controlling hypothermia is essential in anesthesia to limit postoperative complications. Temperature monitoring is therefore essential. However, the reliability of esophageal temperature during open chest lung surgery is discussed and not accurately assessed in the literature.

DETAILED DESCRIPTION:
Controlling hypothermia is essential in anesthesia to limit postoperative complications. Temperature monitoring is therefore essential. However, the reliability of esophageal temperature during open chest lung surgery is discussed and not accurately assessed in the literature.

The investigators therefore decided to evaluate the reliability of the oesophageal temperature in open chest lung surgery by comparing it to the continuous tympanic temperature.

ELIGIBILITY:
Inclusion Criteria:

* all patients needing pulmonary surgery under thoracotomy

Exclusion Criteria:

* patient refusal
* esophageal or otological pathology preventing the installation of thermal probes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults inpatients with thoracotomy surgery, in our University hospital in France
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Correlation between tympanic and oesophageal temperature. | up to 1 day (during the surgery)
  Evaluate the correlation existing between the tympanic temperature, reflection of the central temperature without variation with an open thorax, and oesophageal temperature subject to changes.

SECONDARY OUTCOMES:
Difference of correlation between tympanic and oesophageal temperature during left and right thoracotomy. | up to 1day (during the surgery)
  Evaluate the correlation existing between the tympanic temperature, reflection of the central temperature without variation with an open thorax, and oesophageal temperature subject to changes.

CONTACTS AND LOCATIONS:
Overall Officials: Francis REMERAND, MD-PHD, Study Director — CHU Tours
Locations (2):
- France (2):
  - Department of Anesthesiology - Surgical Intensive Care, University Hospital, Nîmes, Nîmes
  - Department of Anesthesiology - Surgical Intensive Care II, University Hospital, Tours, Tours

REFERENCES:
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Melling AC, Ali B, Scott EM, Leaper DJ. Effects of preoperative warming on the incidence of wound infection after clean surgery: a randomised controlled trial. Lancet. 2001 Sep 15;358(9285):876-80. doi: 10.1016/S0140-6736(01)06071-8. PMID 11567703
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Winkler M, Akca O, Birkenberg B, Hetz H, Scheck T, Arkilic CF, Kabon B, Marker E, Grubl A, Czepan R, Greher M, Goll V, Gottsauner-Wolf F, Kurz A, Sessler DI. Aggressive warming reduces blood loss during hip arthroplasty. Anesth Analg. 2000 Oct;91(4):978-84. doi: 10.1097/00000539-200010000-00039. PMID 11004060
- [Background] Scott AV, Stonemetz JL, Wasey JO, Johnson DJ, Rivers RJ, Koch CG, Frank SM. Compliance with Surgical Care Improvement Project for Body Temperature Management (SCIP Inf-10) Is Associated with Improved Clinical Outcomes. Anesthesiology. 2015 Jul;123(1):116-25. doi: 10.1097/ALN.0000000000000681. PMID 25909970
- [Background] Niven DJ, Gaudet JE, Laupland KB, Mrklas KJ, Roberts DJ, Stelfox HT. Accuracy of peripheral thermometers for estimating temperature: a systematic review and meta-analysis. Ann Intern Med. 2015 Nov 17;163(10):768-77. doi: 10.7326/M15-1150. PMID 26571241
- [Background] Robinson J, Charlton J, Seal R, Spady D, Joffres MR. Oesophageal, rectal, axillary, tympanic and pulmonary artery temperatures during cardiac surgery. Can J Anaesth. 1998 Apr;45(4):317-23. doi: 10.1007/BF03012021. PMID 9597204
- [Background] Gobolos L, Philipp A, Ugocsai P, Foltan M, Thrum A, Miskolczi S, Pousios D, Khawaja S, Budra M, Ohri SK. Reliability of different body temperature measurement sites during aortic surgery. Perfusion. 2014 Jan;29(1):75-81. doi: 10.1177/0267659113497228. Epub 2013 Jul 17. PMID 23863492
- [Background] Rau B, Hunerbein M, Barth C, Schlag PM. [Thoracoscopy is a reliable alternative to thoracotomy in peripheral lung coin lesion]. Langenbecks Arch Chir Suppl Kongressbd. 1997;114:1280-2. German. PMID 9574403
- [Background] Mekjavic IB, Rempel ME. Determination of esophageal probe insertion length based on standing and sitting height. J Appl Physiol (1985). 1990 Jul;69(1):376-9. doi: 10.1152/jappl.1990.69.1.376. PMID 2394660